CLINICAL TRIAL: NCT00928421
Title: An Open-label, Single-dose Pilot Study to Evaluate the Efficacy and Safety of Varisolve® (Polidocanol Endovenous Microfoam) 0.125% [0.2%] for the Treatment of Symptomatic, Visible Varicose Veins With Saphenofemoral Junction (SFJ) Incompetence
Brief Title: An Open-label, Single-dose Pilot Study to Evaluate Varisolve® (Polidocanol Endovenous Microfoam (PEM)) 0.125% [0.2%] for Varicose Veins
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAP.VV014
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Varicose Veins
Keywords: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Varisolve 0.125% (Experimental)
  Interventions: Drug: Polidocanol Endovenous Microfoam 0.125%

INTERVENTIONS:
Drug: Polidocanol Endovenous Microfoam 0.125% — Polidocanol Endovenous Microfoam 0.125%, single dose
  Other Names: Varisolve 0.125%

SUMMARY:
To determine the effect and safety of Varisolve® 0.125% [0.2%]

DETAILED DESCRIPTION:
In patients with SFJ incompetence due to reflux of the Great Saphenous Vein (GSV) or major accessory veins, with venous disease manifested by both symptoms and visible varicosities: using duplex ultrasonography, to evaluate the efficacy of Varisolve® 0.125% [0.2%] as assessed by the elimination of SFJ reflux and/or occlusion of the treated vein

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; age of consent to 75 years
2. Baseline VEINES-Sym Questionnaire score less than 75 points
3. Superficial venous disease manifested by both symptoms and visible varicosities
4. Varicose vein clinical classification CEAP 2 through 5
5. Incompetence of SFJ (reflux > 0.5 seconds on duplex ultrasonography) associated with incompetence of the great saphenous vein (GSV) or other major accessory vein
6. Ability to comprehend and sign an informed consent document and complete study questionnaires in English

Exclusion Criteria:

1. Incompetence of the small saphenous vein (SSV)
2. Ultrasonographic or other evidence of current or previous deep vein thrombosis, occlusion or incompetence
3. Leg obesity impairing the ability to access the vein to be treated and/or to follow the post-procedural compression recommendations.
4. Peripheral arterial disease in the leg to be treated contraindicating post-procedural compression.
5. Reduced mobility (inability to maintain a brisk walk unaided for a minimum of 5 minutes per hour per day).
6. Planned prolonged automobile, bus, or air travel within 4 weeks following treatment, unless the patient can walk for at least 5 consecutive minutes every hour during travel.
7. History of pulmonary embolism or stroke.
8. Major surgery, prolonged hospitalization or pregnancy within 3 months of screening.
9. Current anticoagulation therapy (within 7 days of enrollment).
10. Participation in a clinical study involving an investigational pharmaceutical product or device within the 3 months prior to screening.
11. Previous treatment in this study or in a previous Varisolve® study.
12. Major co-existing disease (e.g. malignancy; pulmonary disease; renal or hepatic insufficiency; serious skin disease/condition that may compromise the ability of the patient to comply with the compression protocol, etc.) or clinically significant laboratory abnormalities.
13. Known allergic response to polidocanol, or severe and multiple allergic reactions.
14. Women of childbearing potential not using effective contraception for at least one month prior to study enrollment and/or unwilling to continue birth control until their last study visit.
15. Pregnant or lactating women.
16. Current alcohol or drug abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Evans, Study Chair — BTG International Inc.
Locations (1):
- Bellevue, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Polidocanol Injectable Foam 0.125%: polidocanol injectable foam 0.125%, single dose
Period: Overall Study
Arm/Group | Polidocanol Injectable Foam 0.125%
Started | 16
Treated With Study Drug | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: all patients treated with polidocanol injectable foam 0.125%
Arm/Group | Polidocanol Injectable Foam 0.125%
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (6.73)

OUTCOME MEASURES:

1. Primary Outcome: Responders to Treatment, Assessed by Duplex Ultrasound
Description: Responders; elimination of reflux through the saphenofemoral junction and/or coplete occlusion of the great saphenous vein at 8 weeks, as measured by duplex ultrasound.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Polidocanol Injectable Foam 0.125%
Number analyzed (Participants) | 16
participants | 9

ADVERSE EVENTS:
Arm/Group | Polidocanol Injectable Foam 0.125%
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 9/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polidocanol Injectable Foam 0.125% (N=16)
extravasation (General disorders) | 1 (1)
local swelling (General disorders) | 2 (2)
limb discomfort (Musculoskeletal and connective tissue disorders) | 8 (8)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No